CLINICAL TRIAL: NCT07077408
Title: iCanCope With NF: Innovating an Efficacious Digital Self-management and Transitional Care Program for Adolescents With Neurofibromatosis
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Hospital for Sick Children (Other)
Collaborators: University Health Network, Toronto (Other)
Responsible Party: Principal Investigator, Jennifer Stinson, Clinician Scientist, The Hospital for Sick Children
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1000081822
Record Dates: First submitted 2025-07-03; First posted 2025-07-22 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2025-07

CONDITIONS: Neurofibromatosis 1
MeSH Terms: conditions — Neurofibromatosis 1

STUDY DESIGN:
Intervention Model Description: A three-arm, parallel group, pilot randomized controlled trial will be conducted.
Masking Description: Blinded data analysis will be conducted by an independent biostatistician
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- iCanCope-NF Youth (Active Comparator): This group will receive access to the intervention on their personal smart phone, or a loaned study phone and charger, for a period of 2 months.
  Interventions: Other: iCanCope-NF Youth app
- iCanCope-NF Youth with Contingency Management (CM) (Experimental): This group (iCanCope+CM) will receive access to the intervention on their personal smart phone, or a loaned study phone, for a period of 2 months. In addition to the standardized orientation and push notifications, this group will also be able to earn incentives aligned with their program engagement.
  Interventions: Other: iCanCope-NF Youth app + CM
- Wait-list control (No Intervention): This group will continue to receive their usual care for 2 months. After completion of their follow-up outcome measures, they will be offered access to the iCanCope-NF Youth program. Participants will be reminded they should us their usual emergency care channels during the study if needed. iCanCope does not replace usual care. If participants need physical or mental health support during the study, they will be directed to resources within their community, primary care provider, specialist, or urgent care/emergency care.

INTERVENTIONS:
Other: iCanCope-NF Youth app — The iCanCope digital app offers symptom tracking, self-management skills training, goal setting, and disease education tailored for neurofibromatosis for youth.
  Arms: iCanCope-NF Youth
Other: iCanCope-NF Youth app + CM — The iCanCope digital app offers symptom tracking, self-management skills training, goal setting, and disease education tailored for neurofibromatosis for youth. In addition to the standardized orientation and push notifications, this app will also allow users to earn incentives aligned with their program engagement.
  Arms: iCanCope-NF Youth with Contingency Management (CM)

SUMMARY:
Neurofibromatosis Type 1 (NF1) often significantly impairs the mental health, social life, self-esteem, and quality of life of adolescent patients. These impacts can be made worse with the experience of NF1-related pain. Nearly three-quarters (73%) of caregivers report that pain interferes with their child's daily functioning, including their mental health, activity, sleep, relationships, and school attendance. Our team has developed the first mobile self-management platform app for adults with NF1-related pain, called iCanCope with NF. It is designed to help people to track their pain, sleep, mood, exercise, and energy level. It helps them set goals, gives suggestions about how to deal with NF1-related pain, and connects them with other individuals living with NF. The goal of this project is to test out a modified version of iCanCope with NF, for youth.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with NF1
* Experience of NF1-related pain or discomfort that interfered with function over the past 2 weeks
* Able to speak and read English

Exclusion Criteria:

* Moderate to severe cognitive impairments that would prevent independent use the iCanCope intervention, as determined through consultation with their health care provider

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2027-03 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Feasibility of iCanCope NF | 8 weeks
  Success will be defined as meeting the following four combined criteria: 1) accrual rate >70% 2) attrition rate <20%; 3) technical difficulties in fewer than 10% of cases; and acceptability of mean 4 or higher on the acceptability e-scale.

SECONDARY OUTCOMES:
Pain Interference | 8 weeks
  measured by the 16-item Pain Impact Scale from the PedsQL NF1 module. This measures reflect how much pain hinders activity and functioning.
Pain Severity | 8 weeks
  Pain severity will be measured using the 6-item validated Pain Scale from the PedsQL NF1 module.
Pain management | 8 weeks
  Pain management is assessed will be measured using the 2-item validated Pain Management Scale from the PedsQL NF1 module
Depressive symptoms | 8 weeks
  Depressive symptoms will be measured using the validated 8-item Patient-Reported Outcomes Measurement Information System (PROMIS®) Depression Short form for the assessment of depressive symptoms.
Anxiety | 8 weeks
  Anxiety will be assessed using the validated 10-item Worry Scale from the PedsQL NF1 Module.
Transition readiness | 8 weeks
  Transition readiness which examines how prepared a pediatric patient is for adult care. This will be assessed using the 20-item validated Transition Readiness Assessment Questionnaire Version 5 (TRAQ 5.0)
Health-related quality of life | 8 weeks
  Health-related quality of life will be measured using the 23-item PedsQL 4.0 Generic49 questionnaire.

IPD SHARING:
Plan to Share IPD: No